CLINICAL TRIAL: NCT04063345
Title: A Prospective, Open Label, Multicenter and Randomized Study of Clinical Outcomes of Intravascular Ultrasound -Guided and Angiography-Guided Primary Percutaneous Intervention in Patients With Acute ST Segment Elevated Myocardial Infarction
Brief Title: Long-term Clinical Outcomes of intraVascular Ultrasound-guided vs Angiography-guided Primary pErcutaneous Intervention in Patients With Acute ST Segment Elevated Myocardial Infarction
Acronym: LOVEinSTEMI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo No. 1 Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Shanghai Chest Hospital (Other); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT015
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI; Intravascular ultrasound; Angiography; Primary percutaneous intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS-guided PCI (Experimental): Percutaneous intervention under IVUS-guidance
  Interventions: Procedure: IVUS-guided PCI
- Angiography-guided PCI (Active Comparator): Percutaneous intervention under angiograhy-guidance only
  Interventions: Procedure: Angiography-guided PCI

INTERVENTIONS:
Procedure: IVUS-guided PCI — Performing intravascular ultrasound before or/and after percutaneous intervention
  Arms: IVUS-guided PCI
Procedure: Angiography-guided PCI — Performing percutaneous intervention without intravascular ultrasound guidance
  Arms: Angiography-guided PCI

SUMMARY:
To examine the impact of IVUS guidance on clinical outcomes in the patient with Acute ST Segment Elevated Myocardial Infarction.

DETAILED DESCRIPTION:
Intravascular ultrasound (IVUS) has been increasingly used as a guide for percutaneous coronary intervention (PCI) during elective as well as emergent clinical scenario. Recent small number randomized studies, large scale registries as well as meta-analysis have consistently demonstrated advantages of IVUS-guidance over angiography-guide alone with respect to the lower incident of death, myocardial infarction and target vessel revascularization.

There are sparse data available on the clinical impact of IVUS-guided PCI in the setting of acute myocardial infarction (AMI) and its use remains a matter of controversy as shown by previous studies. This study is to examine the impact of IVUS guidance on clinical outcomes in the patient with Acute ST Segment Elevated Myocardial Infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical inclusion criteria:

  1. Age > 18 years
  2. Onset of STEMI > 30 minutes, but < 12 hours
  3. ST segment elevation in at least 2 contiguous leads of≥ 1mm or newly developed LBBB on ECG
  4. Willing and able to provide informed consent
* Angiographic inclusion criteria:

  1. Having at least one infarct-related coronary artery, of which (1) the Culprit lesion is suitable for stenting (2) the reference diameter of culprit vessel is ≥ 2.5 mm but ≤ 4 mm (3) the TIMI flow is ≤ 1 in culprit lesion segment prior to guide wire crossing
  2. No excessive tortuosity and calcification in the culprit lesion segment that allowing stent implantation

Exclusion Criteria:

* Clinical exclusion criteria:

  1. Contraindicating to any concomitant study medications
  2. Having cardiogenic shock with hemodynamic instability
  3. A history of bleeding diathesis or known coagulopathy
  4. A history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months; or a history of intracranial tumor, aneurysm or arteriovenous malformations; or a history of active peptic ulcer or active gastrointestinal (GI) bleeding within the past 2 months; or planned major procedure within 6 weeks; or known platelet count < 100,000 /mm3 or Hb < 10 g/dL
  5. Planned surgery which may cause discontinuation of ADP-receptor antagonist
  6. Other serious illness (e.g., cancer) that may reduce life expectancy to less than 1 year
  7. Repeated MI within 7 days of hospitalization for acute MI
* Anigographic Exclusion Criteria:

  1. Bifurcated lesion unable to identify the culprit lesion
  2. The culprit lesion is located in the left main artery
  3. Diffusive lesions without distinguishable culprit lesion
  4. Previous stent implantation in the culprit lesion segment or STEMI caused by stent thrombosis
  5. Likely CABG procedure within 30 days
  6. Renal failure requiring or during dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) rate | 1 year
  Defined as cardiac death, myocardial infarction (MI, Q-wave and non-Q-wave) and target vessel revascularization (TVR)

SECONDARY OUTCOMES:
MACE rate | 2-3 years
Target lesion revascularization (TLR) rate | 2-3 years
Target lesion failure (TLF) rate | 2-3 years
TVR rate | 2-3 years
Target vessel failure (TVF) rate | 2-3 years
MI (Q-wave and non-Q-wave) rat | 2-3 years
Cardiac death rate | 2-3 years
Non-cardiac death rate | 2-3 years
All death (cardiac and non-cardiovascular) rate | 2-3 years
Stent Thrombosis (ST) rate (ARC definite/probable) | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD, PhD, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China